CLINICAL TRIAL: NCT03952403
Title: A Three Arm, Randomized, Double-Blind, Multicenter, Phase 3 Study of HLX10(Anti-PD-1 Antibody) in Combination With Carboplatin Plus (+) Pemetrexed With or Without HLX04(Avastin Biosimilar) Compared With Carboplatin+Pemetrexed in 1L Stage IIIB/IIIC or IV Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of HLX10 in Combination With Carboplatin Plus (+) Pemetrexed With or Without HLX04 Compared With Carboplatin+Pemetrexed in 1L Advanced Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-002-NSCLC301
Record Dates: First submitted 2019-05-06; First posted 2019-05-16 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma; Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma | interventions — Carboplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1-Cohort 1 (HLX10+HLX04+Carboplatin+Pemetrexed) (Experimental): Participants will receive IV infusion of HLX10 and HLX04 on Day 1 of each 21-day cycle followed by IV infusion of Carboplatin and Pemetrexed on Day 1 of each 21-day cycle for 4 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants will receive IV infusion of HLX10 until loss of clinical benefit and HLX04 and Pemetrexed until progressive disease, unacceptable toxicity, or death during maintenance treatment phase.
  Interventions: Drug: HLX10, an engineered anti-PD-1 antibody; Drug: HLX04, a bevacizumab biosimilar; Drug: Carboplatin; Drug: Pemetrexed
- Part 2-Arm A (HLX10+HLX04+Carboplatin+Pemetrexed) (Experimental): Participants will receive IV infusion of HLX10 and HLX04 on Day 1 of each 21-day cycle followed by IV infusion of Carboplatin and Pemetrexed on Day 1 of each 21-day cycle for 4 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants will receive IV infusion of HLX10 until loss of clinical benefit and HLX04 and Pemetrexed until progressive disease, unacceptable toxicity, or death during maintenance treatment phase.
  Interventions: Drug: HLX10, an engineered anti-PD-1 antibody; Drug: HLX04, a bevacizumab biosimilar; Drug: Carboplatin; Drug: Pemetrexed
- Part 2-Arm B (HLX10+HLX04 placebo+Carboplatin+Pemetrexed) (Experimental): Participants will receive IV infusion of HLX10 and HLX04 placebo on Day 1 of each 21-day cycle followed by IV infusion of Carboplatin and Pemetrexed on Day 1 of each 21-day cycle for 4 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants will receive IV infusion of HLX10 until loss of clinical benefit and Pemetrexed until progressive disease, unacceptable toxicity, or death during maintenance treatment phase.
  Interventions: Drug: HLX10, an engineered anti-PD-1 antibody; Drug: Carboplatin; Drug: Pemetrexed
- Part 2-Arm C (HLX10 placebo+HLX04 placebo+Carboplatin+Pemetrexed) (Active Comparator): Participants will receive IV infusion of HLX10 placebo and HLX04 placebo on Day 1 of each 21-day cycle followed by IV infusion of Carboplatin and Pemetrexed on Day 1 of each 21-day cycle for 4 cycles or until loss of clinical benefit whichever occurs first, during induction treatment phase. Participants will receive IV infusion Pemetrexed until progressive disease, unacceptable toxicity, or death during maintenance treatment phase.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: HLX10, an engineered anti-PD-1 antibody — HLX10 will be administered as IV infusion at a dose of 4.5mg/kg on Day 1 of each 21-day cycle until loss of clinical benefit or up to 2 year.
  Arms: Part 1-Cohort 1 (HLX10+HLX04+Carboplatin+Pemetrexed); Part 2-Arm A (HLX10+HLX04+Carboplatin+Pemetrexed); Part 2-Arm B (HLX10+HLX04 placebo+Carboplatin+Pemetrexed)
Drug: HLX04, a bevacizumab biosimilar — HLX04 will be administered as IV infusion at a dose of 15 milligrams per kilogram (mg/kg) on Day 1 of each 21-day cycle until progressive disease, unacceptable toxicity, death or up to 2 year.
  Arms: Part 1-Cohort 1 (HLX10+HLX04+Carboplatin+Pemetrexed); Part 2-Arm A (HLX10+HLX04+Carboplatin+Pemetrexed)
Drug: Carboplatin — Carboplatin will be administered at area under the concentration-time curve (AUC) 5 on Day 1 of each 21-day cycle for 4 cycles, or until loss of clinical benefit whichever occurs first.
Drug: Pemetrexed — Pemetrexed will be administered as IV infusion at a dose of 500 milligrams per square meter (mg/m2) on Day 1 of each 21-day cycle until progressive disease, unacceptable toxicity, death or up to 2 year.

SUMMARY:
This study involves a two-part design. Part 1 is designed to evaluate the safety and tolerability of the 4 drug (HLX10+HLX04+carboplatin+pemetrexed). Part 2 is a randomized, open-label study, which will evaluate the safety and efficacy of HLX10 in combination with carboplatin+pemetrexed with or without HLX04(biosimilar of avastin) compared with treatment with carboplatin+pemetrexed in 1st line Stage IIIB/IIIC or IV non-squamous NSCLC. Participants will be randomized in a 1:1:1 ratio to Arm A (HLX10+HLX04+Carboplatin+Pemetrexed), Arm B (HLX10+HLX04 placebo+Carboplatin+Pemetrexed), or Arm C (HLX10 placebo + HLX04 placebo+Carboplatin+Pemetrexed).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, Stage IIIB/IIIC or IV non-squamous NSCLC
2. Participants with no EGFR, ALK and ROS1 mutation.
3. Participants with no prior treatment for Stage IIIB/IIIC or IV non-squamous NSCLC
4. Measurable disease as defined by RECIST v1.1
5. Eastern Cooperative Oncology Group performance status 0 or 1
6. Adequate hematologic and end organ function

Exclusion Criteria:

1. Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
2. Active central nervous system metastases
3. Prior treatment with cluster of differentiation immune checkpoint blockade therapies or Bevacizumab
4. Has received a surgical operation within 4 weeks from the initial drug administration
5. Active or suspected autoimmune diseases. Subjects in a stable state with no need for systemic immunosuppressant therapy are allowed to enroll.
6. Currently having or have had interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis and severe impaired pulmonary function that may interfere with the detection and management of suspected drug-related pulmonary toxicity
7. Any active infection requiring systemic anti-infective therapy within 14 days prior to study drug administration
8. Uncontrollable active infection(s)
9. History of immunodeficiency, including HIV antibody positive
10. active hepatitis B; or hepatitis C virus infections
11. Has bleeding tendency
12. History of severe cardiovascular diseases
13. Known gastrointestinal diseases as follows, Gastrointestinal perforation, abdominal fistula or abdominal abscess within 6 months before signing the informed consent; History of poorly controlled or recurrent inflammatory bowel disease; Active peptic ulcers, or > moderate esophageal varices
14. Pregnant or breastfeeding female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Part 1 Safety and tolerability of study treatment | baseline to 21 days
Part 2-Progression Free Survival (PFS) as Determined by the IRRC using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Baseline until disease progression or death, whichever occurs first (up to approximately 24months)

SECONDARY OUTCOMES:
Part 2-Overall survival (OS), as a major secondary endpoint | Baseline until death (up to approximately 36 months)
Part 1 and 2-Incidence rates of AEs and SAEs | Baseline up to approximately 36months
Part 1-Overall survival (OS) | Baseline up to approximately 36months
Part 1 and Part 2-PFS (assessed by the investigator according to RECIST v1.1) in Part 1 and 2; PFS (assessed by IRRC according to RECIST v1.1) in Part 1 | Baseline until disease progression or death, whichever occurs first (up to approximately 36months)
Part 1 and 2-Objective response rate (ORR, assessed by IRRC and investigator according to RECIST v1.1 criteria) | Baseline up to approximately 36 months
Part 1 and 2-Duration of response (DOR, assessed by IRRC and investigator according to RECIST v1.1 criteria) | Baseline up to approximately 36 months
Part 2-PFS2 (assessed by IRRC) | Baseline up to approximately 36months
Part 1 and 2-Pharmacokinetics (PK): serum HLX10 concentration | Baseline up to approximately 36 months
Part 1 and 2-Immunogenicity evaluation: positive anti-drug antibody (ADA) rate | Baseline up to approximately 36 months
Part 1 and 2-PD-L1 expression level | Baseline
Part 1 and 2-Microsatellite instability(MSI) | Baseline
Part 1 and 2-Tumor mutation burden(TMB) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yankai Shi, professor, Principal Investigator — Cancer Hospital Chinese Academy of Medical Sciences (CAMS)
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences (CAMS), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang L, Hao X, Hao Y, Hu Y, Chen C, Chen B, Huang Y, Zang A, Wang Y, Chen Z, Zhuang W, Shi J, Ren X, Nie L, Yu G, Luo F, Mao Y, Wang X, Li B, Bai Y, Shi J, Ni H, Yu H, Li J, Wang Q, Zhu J, Shi Y; ASTRUM-002 Study Group. First-line serplulimab plus chemotherapy with or without HLX04 versus chemotherapy in locally advanced or metastatic non-squamous non-small-cell lung cancer (ASTRUM-002): a randomised, double-blind, multicentre phase 3 trial. Lancet Respir Med. 2025 Dec 4:S2213-2600(25)00263-2. doi: 10.1016/S2213-2600(25)00263-2. Online ahead of print. PMID 41354044
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107